CLINICAL TRIAL: NCT06754501
Title: A Phase 2 Clinical Trial Evaluating the Efficacy and Safety of Dual Immune Checkpoint Inhibition With Anti-PD-L1 (Atezolizumab) and Anti-TIGIT (Tiragolumab) in Cancer of Unknown Primary
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Strategic Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0210; NCI-2024-10697 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2024-12-30; First posted 2024-12-31 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — atezolizumab; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Atezolizumab + Tiragolumab (Experimental)
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — Given by vein
Drug: Tiragolumab — Given by vein

SUMMARY:
The goal of this clinical research study is to learn if the combination of atezolizumab and tiragolumab can help to control cancers of unknown primary. The safety and effects of this drug combination will also be studied

DETAILED DESCRIPTION:
Primary Objectives:

To assess the anti-tumor activity of tiragolumab and atezolizumab in patients with CUP.

Primary Endpoint: confirmed ORR as per RECISTv1.1.

Secondary Objectives:

To assess the best objective response rate (ORR) (investigator assessed), disease control rate (DCR), duration of response (DOR), progression-free survival (PFS) overall survival (OS) in patients with CUP.

Secondary Endpoints: Best overall response rate per RECISTv1.1 (investigator assessed), DCR, DOR, PFS, and OS

ELIGIBILITY:
Inclusion Criteria:

● Patients must have histopathological confirmed unresected, locally advanced, recurrent, or metastatic CUP. Patients must have undergone standard work-up to attempt to find the primary tumor prior to enrollment.

Patients must be refractory or intolerant to at least one line of systemic chemotherapy or ineligible for cytotoxic chemotherapy.

* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for nonnodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of tiragolumab in combination with atezolizumab in patients <18 years of age, children are excluded from this study.
* ECOG performance status of 0-1.
* Patients must have adequate organ and marrow function as defined below:

  * ANC > 1.5 x 109 /L (1500/L) without granulocyte colony-stimulating factor support.
  * Lymphocyte count > 0.5 x 109 /L (500/L).
  * Platelet count > 100 x 109 /L (100,000/L) without transfusion.
  * Hemoglobin > 90 g/L (9 g/dL).
  * Patients may be transfused to meet this criterion.
  * AST, ALT, and ALP < 2.5 x upper limit of normal (ULN).
  * Total bilirubin < 1.5 x ULN with the following exception:
  * Patients with known Gilbert disease: total bilirubin < 3 x ULN.
  * Creatinine clearance > 45 mL/min (calculated using the Cockcroft-Gault formula).
  * Serum albumin > 25 g/L (2.5 g/dL).
  * For patients not receiving therapeutic anticoagulation: INR and aPTT < 1.5 x ULN.
  * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen.

Is able to provide archival or fresh tissues for correlative analysis with obtainable results.

* Negative HIV test at screening with the following exception: individuals with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4+ T cell count > 200/L, and have an undetectable viral load.
* Negative hepatitis B surface antigen (HBsAg) test at screening
* Positive hepatitis B surface antibody (HBsAb) test at screening, or negative HBsAb at screening accompanied by either of the following:

  * Negative total hepatitis B core antibody (HBcAb).
  * Positive total HBcAb test followed by quantitative hepatitis B virus (HBV) DNA < 500 IU/mL.
  * The HBV DNA test will be performed only for patients who have a negative HBsAg test, a negative HBsAb test, and a positive total HBcAb test.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening

  - The HCV RNA test will be performed only for patients who have a positive HCV antibody test.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.

Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.

* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Patients who are pregnant or breastfeeding.
* Ability to understand and the willingness to sign a written informed consent document.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception:

  * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 90 days after the final dose of tiragolumab, 5 months after the final dose of atezolizumab.
  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (> 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Per this definition, a woman with a tubal ligation is considered to be of childbearing potential. The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.

The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

* With a female partner of childbearing potential, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period, for 90 days after the final dose of tiragolumab. Men must refrain from donating sperm during this same period.
* With a pregnant female partner, men must remain abstinent or use a condom during the treatment period for 90 days after the final dose of tiragolumab, and per the requirements of local label after the final dose of paclitaxel, pemetrexed, gemcitabine, carboplatin, or cisplatin to avoid exposing the embryo.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.

For Cohort A: Patients should have BostonGene Tumor Portrait testing that demonstrates either Immune-Enriched (IE/F) or Immune-Enriched, Non-Fibrotic (IE) subtypes.

● For Cohort B: Patients should have BostonGene Tumor Portrait testing that demonstrates either Fibrotic (F) or Desert (D) subtypes.

Exclusion Criteria:

* Patients who have received treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, LAG-3inhibitor, or anti-CTLA-4 antibody, or any other antibody or drug that specifically targets Tcell co-stimulation or immune checkpoint pathways.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e.,have residual toxicities > NCI CTCAE v5.0 Grade 1) with the exception of alopecia, events that are not clinically significant, or asymptomatic laboratory abnormalities.
* Patients who are receiving any other investigational agents.
* History of leptomeningeal disease
* Uncontrolled tumor-related pain

  * Patients requiring pain medication must be on a stable regimen at study entry.
  * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
  * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Patients with indwelling catheters (e.g., PleurX) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium <12 mg/dL or corrected serum calcium > ULN)

Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the exceptions listed below:

Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study. Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.

Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

* Rash must cover < 10% of body surface area.
* Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
* 'There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.

  * History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
  * Active tuberculosis Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
  * Patients who are taking prohibited medications as detailed in Appendix A.
  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
  * Patients with psychiatric illness/social situations that would limit compliance with study requirements.
  * History of malignancy other than cancer of unknown primary within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
  * Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia, or any active infection that could impact patient safety
  * Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment

    - Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
  * Patients with a history of uncontrolled auto-immune disorders requiring systemic immunosuppression.
  * Has undergone major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment or is scheduled to receive major surgery during the course of the trial.
  * Has an active or poorly controlled serious infections.
  * Has symptomatic congestive heart failure (NYHA Class II-IV) or symptomatic or poorly controlled arrhythmia.
  * Has a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
  * Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during study treatment, within 90 days after the final dose of tiragolumab, or within 5 months after the final dose of atezolizumab
  * Positive Epstein-Barr virus (EBV) viral capsid antigen immunoglobulin M (IgM) test at screening

    - An EBV polymerase chain reaction (PCR) test should be performed as clinically indicated to screen for acute infection or suspected chronic active infection. Patients with a positive EBV PCR test are excluded.
  * Had any arterial thromboembolic event within 6 months prior to enrollment, including myocardial infarction, unstable angina, cerebrovascular accident, or transient cerebral ischemic attack.
  * Has a history of clinically significant deep venous thrombosis, pulmonary embolism, or other serious thromboembolic events within 3 months prior to enrollment (having an implantable port or catheter-related thrombosis or incidental pulmonary embolism detected on scan without symptoms or superficial venous thrombosis is not considered to be a "serious" thromboembolisms).

Has significant malnutrition, such as those requiring continuous parenteral nutrition ≥7 days.

Allowed are those who received intravenous treatment for malnutrition that ended more than 4 weeks before the first dose of study treatment.

* Has hepatic encephalopathy, hepatorenal syndrome, or cirrhosis with Child-Pugh Class B or C.
* Has bowel obstruction or history of any of the following diseases: inflammatory bowel disease, extensive bowel resection (partial colectomy or extensive small intestine resection accompanied with chronic diarrhea), Crohn's disease, or ulcerative colitis.
* Has an acute or chronic diseases, psychiatric disorders, or laboratory abnormality that may lead to the following consequences: increased investigational drug-related risks, or interference with interpretation of trial results, or is otherwise considered ineligible for participating in the trial by the investigators.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and IL-2) within 4 weeks or 5 drug-elimination half-lives (whichever is longer) prior to initiation of study treatment.

Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor- [TNF-] agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

* Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
* Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.

  * Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or tiragolumab formulation.
  * Known allergy or hypersensitivity to any component of the chemotherapy regimen the patient may receive during the study
  * Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment, within 90 days after the final dose of tiragolumab or 5 months after the final dose of atezolizumab.
* Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

  * Patients may not concomitantly use any of the prohibited therapies detailed in Appendix A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Huey, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org